CLINICAL TRIAL: NCT00611754
Title: Phase II Study of Oxaliplatin in Combination With 5-Fluorouracil (5-FU) in 1st Line Treatment of Locally Advanced or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Phase II Study of Oxaliplatin in Combination With 5-Fu in 1st Line Treatment of Locally Advanced or Metastatic Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Nathalie Billon/Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFC_7276
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-01

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Oxaliplatin; Fluorouracil

INTERVENTIONS:
Drug: Oxaliplatin, 5-FU — Oxaliplatin: 130 mg/m² in 500 mL of 5% glucose solution as a 2-hour intravenous (IV) infusion on Day 1 and repeated every 3 weeks; 5-FU: following oxaliplatin administration, 1000 mg/m²/day as a continuous IV infusion from Day 1 toDay 4, every 3 weeks.Dose adjustments were made if the patient experienced AEs.
  Other Names: Eloxatin®, Fluorouracil

SUMMARY:
To evaluate the efficacy of first line oxaliplatin in combination with 5-fluorouracil (5-FU) in patients with advanced inoperable or metastatic head and neck cancer and to investigate the safety profile of this regimen in the above indication and consider other criteria of efficacy (clinical benefit, survival)

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-70 years, with inoperable locally advanced or metastatic squamous cell carcinoma of the head and neck (stage III-IV) histologically proven, no prior chemo and/or hormone therapy for metastatic disease or local recurrence (adjuvant or neo-adjuvant chemotherapy or radio-chemotherapy was allowed if finished since more than 6 months before inclusion and cisplatinum total dose used < or=to 300 mg/m² or carboplatinum total dose used < or=to 200mg/m²), at least 1 target lesion (measurable in 2 dimensions > or=to 20 mm on computed tomography (CT) or magnetic resonance imaging (MRI) evaluated < 15 days before start of study treatment, outside of irradiated fields),performance status (PS) < or =to 2 World Health Organization (WHO), weight loss < 5% normal weight,hemoglobin > or =to 10 g/dL, neutrophils > or =to 2000/mm3, platelets > or =to 100,000/mm3 , creatinine < or =to 1.5 x upper limit of normal (ULN), bilirubin < or =to .5 x ULN, alanine amino-transferase (ALT)/aspartate amino-transferase (AST)< or =to 2.5 x ULN (5 x ULN if liver metastases), clotting: prothrombin time (PT) > or =to 60%. Written informed consent signed by patient and doctor prior to all study procedures -

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2000-05; Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of first line oxaliplatin in combination with 5-fluorouracil (5-FU) in patients with advanced inoperable or metastatic head and neck cancer.

SECONDARY OUTCOMES:
To investigate the safety profile of this regimen in the above indication and consider other criteria of efficacy (clinical benefit, survival)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Billon, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Paris, France